CLINICAL TRIAL: NCT05906199
Title: A Prospective, Randomized, Active-controlled, Parallel, Open, Multi-center, Phase IV, Exploratory Clinical Trial to Compare the Effects of Improving the Carotid Artery Intima Media Thickness and Changing Lipid Levels by Cilostazol/Ginkgo Leaf Extract (Renexin CR) and Aspirin (Aspirin Protect Tab.) in Diabetic Peripheral Angiopathy.
Brief Title: A Study to Compare the Effects of Improving the Carotid Artery Intima Media Thickness and Changing Lipid Levels by Cilostazol/Ginkgo Leaf Extract and Aspirin in Diabetic Peripheral Angiopathy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNX_001
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Peripheral Angiopathy
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Renexin CR 200/160mg (Experimental): Single oral administration of Renexin CR 200/160mg, QD
  Interventions: Drug: Renexin CR 200/160mg
- Aspirin 100mg (Active Comparator): Single oral administration of Aspirin 100mg, QD
  Interventions: Drug: Aspirin 100mg

INTERVENTIONS:
Drug: Renexin CR 200/160mg — Single oral administration of Renexin CR 200/160mg, QD
  Other Names: Renexin CR
  Arms: Renexin CR 200/160mg
Drug: Aspirin 100mg — Single oral administration of Aspirin 100mg, QD
  Other Names: Aspirin
  Arms: Aspirin 100mg

SUMMARY:
This study is to compare and evaluate the effect of improving the carotid IMT and lipid level of the Cilostazol/Ginkgo leaf extract group with the aspirin administrated group in patients with diabetic peripheral angiopathy.

DETAILED DESCRIPTION:
A Prospective, Randomized, Active-controlled, Parallel, Open, Multi-center, Phase IV

ELIGIBILITY:
<Inclusion Criteria>

1. Male or female aged between 20 years and 75 years(inclusive)
2. Patients who diagnosed as type 2 diabetes and diabetic peripheral angiopathy
3. Patients with a maximum intra-carotid membrane thickness (maximum IMT) of 0.9 mm or more among the thickest areas, including plaques, in the CCA, ICA, and Bulb three areas of the carotid artery

<Exclusion Criteria>

1. Patients who diagnosed with type 1 diabetes, secondary diabetes, or gestational diabetes
2. Patients with cerebrovascular or cardiovascular complications within 6 months of screening (cerebral infarction, transient ischemic seizures, myocardial infarction, unstable angina, coronary artery bypass graft(CABG), PCI, etc.)
3. Patients with bleeding (hemophilia, capillary weakness, intracranial hemorrhage, upper digestive tract hemorrhage, urinary tract hemorrhage, hematopoietic hemorrhage, active digestive ulcers, etc.) or peptic ulcers within 3 months of screening
4. Patient who took anticoagulants, antiplatelet drugs including aspirin, cilostazol, thrombolytic agents, prostaglandin E1 and glucagon-like peptide -1 (GLP-1) receptor agonist within 2 weeks of the baseline

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Changes in carotid IMT | 24weeks, 48weeks
  Changes in carotid IMT after 24weeks, 48weeks of administration compared to before administration of investigational product

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - SKChemicals, Seongnam, Gyunggi-do
  - SK chemicals, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang YC, Kim MK, Park JH, Yun HM, Kim SY, Lim S. Comparison of Efficacy and Safety of Cilostazol/Extract of Ginkgo biloba vs. Aspirin in Carotid Atherosclerosis in Patients with Diabetes Mellitus. Diabetes Metab J. 2025 Aug 13. doi: 10.4093/dmj.2025.0146. Online ahead of print. PMID 40803668